CLINICAL TRIAL: NCT06322394
Title: A Multicentre, Randomised, Double-blind, Placebo-parallel Controlled Phase II Clinical Trial Evaluating the Efficacy and Safety of BXOS110 Injection in the Treatment of Acute Ischaemic Stroke Within 3 Hours of Onset
Brief Title: BXOS110 Injection in the Treatment of Acute Ischaemic Stroke
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biocells (Beijing) Biotech Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BXOS110-Ⅱ-2023-12
Record Dates: First submitted 2024-03-12; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BXOS110 high-dose group (Experimental): Name:BXOS110 Dosage form:injection Dosage:3.0 mg/kg, maximum dose not exceeding 300 mg Frequency:Frequency of injection is once Duration:10±1 min
  Interventions: Drug: high-dose BXOS110
- BXOS110 low-dose group (Experimental): Name:BXOS110 Dosage form:injection Dosage:2.0 mg/kg, maximum dose not exceeding 300 mg Frequency:Frequency of injection is once Duration:10±1 min
  Interventions: Drug: low-dose BXOS110
- Placebo control group (Placebo Comparator): Dosage:0 mg/kg Frequency:Frequency of injection is once Duration:10±1 min
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: high-dose BXOS110 — 3.0 mg/kg, maximum dose not exceeding 300 mg，Participants received one administration by intravenous infusion.
  Other Names: BXOS110
  Arms: BXOS110 high-dose group
Drug: low-dose BXOS110 — 2.0 mg/kg, maximum dose not exceeding 200 mg，Participants received one administration by intravenous infusion.
  Other Names: BXOS110
  Arms: BXOS110 low-dose group
Drug: Placebo — Does not contain any test drug active ingredients，Participants received one administration by intravenous infusion.
  Arms: Placebo control group

SUMMARY:
The purpose of this study was to evaluate the effectiveness of early administration of BXOS110 for injection in reducing overall disability in patients with acute ischaemic stroke.

DETAILED DESCRIPTION:
This trial was conducted in a multicentre, randomised, double-blind, placebo-parallel controlled design, with a total of three groups of 100 subjects in each of the three planned groups, namely, the BXOS110 high-dose group (3.0 mg/kg, with a maximum dose of up to 300 mg), the BXOS110 low-dose group (2.0 mg/kg, with a maximum dose of up to 200 mg) and the placebo-control group, with the aim of exploring the efficacy and safety of BXOS110 at different doses of BXOS110. efficacy and safety of BXOS110.

The trial was divided into a screening/baseline period, a treatment period and a follow-up period. In the screening/baseline phase, patients signed an informed consent form within 3 hours of stroke onset to enter the trial, and after completing the screening and procedures related to the trial, subjects who met the enrolment requirements were randomly assigned to the BXOS110 high-dose group, the BXOS110 low-dose group, or a placebo-controlled group in a ratio of 1: 1: 1. During the treatment phase, subjects were randomly grouped into groups to start the intravenous treatment, and evaluations were carried out immediately after the administration of BXOS110. immediately after administration; during the Follow-up Period, subjects were evaluated for effectiveness and safety on Day 2, Day 3, Day 10, or at discharge (whichever occurred earlier), Day 30, and Day 90 after administration.

ELIGIBILITY:
Inclusion Criteria:

1. Age18~85 (including 18 and 85 years)，no gender limitation;
2. Subjects diagnosed with acute ischaemic stroke according to the Chinese Guidelines for Clinical Management of Cerebrovascular Disease (2nd edition);
3. 6 ≤ NIHSS score ≤ 20 before randomisation;
4. Within 3h of stroke onset and expected to be able to start receiving the investigational product within 3 h of stroke onset (note: stroke onset time was calculated from the onset time of stroke symptoms; if stroke onset occurs during sleep, the stroke onset time should be taken as the latest normal appearance time);
5. First stroke onset, or have a history of stroke but good prognosis (mRS score ≤1);
6. Subjects who are able to understand and comply with the study procedures, and who agree to sign the study informed consent form in writing to indicate that they are willing to participate in the trial (the informed consent form can be signed by subjects or their legal representatives).

Exclusion Criteria:

1. Imaging confirmed intracranial hemorrhagic disease (hemorrhagic stroke, epidural hematoma, intracranial hematoma, subarachnoid hemorrhage, ventricular hemorrhage, traumatic cerebral hemorrhage, etc.);
2. Severe disturbance of consciousness: NIHSS 1a score ≥2 points;
3. After aggressive antihypertensive therapy, hypertension still not under control: systolic blood pressure ≥180 mmHg, or diastolic blood pressure ≥110 mmHg;
4. Severe hyperglycemia/hypoglycemia: blood glucose≥400 mg/dL (22.2 mmol/L), or ≤50 mg/dL (2.8 mmol/L);
5. Heart rate < 50 beats /min or heart rate > 120 beats /min; Heart failure, unstable angina pectoris, acute myocardial infarction, and severe arrhythmias within the previous 6 months, as determined by the investigators to be severe heart disease, affected participants;
6. Previously diagnosed severe hepatic and renal dysfunction and determined by the investigators as affect the subjects;
7. Patients who have been treated with neuroprotective agents after current stoke onset;
8. Have a epilepsy history or have epilepsy symptoms after current stoke onset;
9. Combined with other mental illnesses, resulting in inability or unwillingness to cooperate;
10. Combined with claudication, osteoarthropathy, etc., resulting in limb movement dysfunction, which is determined by investigators to affect neurological function test;
11. History of severe head trauma or stroke within 3 months before screening;
12. History of severe food or drug allergy, or known allergy to the investigational drug and its excipients;
13. Expected survival period is less than 3 months;
14. Pregnant, planning pregnancy or breastfeeding patients;
15. Suspected or confirmed history of alcohol or drug abuse;
16. Participated in other drug or device clinical trial within the 3 months prior to screening or are participating in a other clinical trial;
17. Other conditions, and the investigator assessed that participation in the study might increase the patient's risk or that participation in the study was deemed inappropriate by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with mRS score 0-2 on day 90 | Day 90
  Modified Rankin scale The Rankin scale was devised in 1957 for assessment of stroke outcomes, and was modified in 1988 to improve its comprehensiveness.The modified version, or mRS, has since been commonly used to assess disability after a stroke.
  The mRS attempts to measure functional independence, incorporating the WHO components of body function, activity, and participation. The scale is defined categorically with seven different grades: 0 indicates no symptoms, 5 indicates severe disability, and 6 indicates death.
  A 1-point shift on this scale is often deemed clinically significant because of the large category sizes. Patients may use adaptive devices and still be considered independent, but the need for supervision or even minimum aid from another person is scored as dependent.

SECONDARY OUTCOMES:
Proportion of subjects with mRS score 0-1 on day 90 | Day 90
  The modified version, or mRS, has since been commonly used to assess disability after a stroke.
  The mRS attempts to measure functional independence, incorporating the WHO components of body function, activity, and participation. The scale is defined categorically with seven different grades: 0 indicates no symptoms, 5 indicates severe disability, and 6 indicates death.
  A 1-point shift on this scale is often deemed clinically significant because of the large category sizes. Patients may use adaptive devices and still be considered independent, but the need for supervision or even minimum aid from another person is scored as dependent.
Day 90 mRS Displacement Analysis | Day 90
  The modified version, or mRS, has since been commonly used to assess disability after a stroke.
  The mRS attempts to measure functional independence, incorporating the WHO components of body function, activity, and participation. The scale is defined categorically with seven different grades: 0 indicates no symptoms, 5 indicates severe disability, and 6 indicates death.
  A 1-point shift on this scale is often deemed clinically significant because of the large category sizes. Patients may use adaptive devices and still be considered independent, but the need for supervision or even minimum aid from another person is scored as dependent.
Proportion of subjects with NIHSS scores ≤1 on day 10 (or at discharge) | Day 10
  The NIHSS is a 15-item impairment scale, which provides a quantitative measure of key components of a standard neurological examination.
  The scale assesses level of consciousness, extraocular movements, visual fields, facial muscle function, extremity strength, sensory function, coordination (ataxia), language (aphasia), speech (dysarthria), and hemi-inattention (neglect).
Proportion of subjects with a ≥4-point reduction in NIHSS score from baseline at day 10 (or at discharge) | D10
  The NIHSS is a 15-item impairment scale, which provides a quantitative measure of key components of a standard neurological examination.
  The scale assesses level of consciousness, extraocular movements, visual fields, facial muscle function, extremity strength, sensory function, coordination (ataxia), language (aphasia), speech (dysarthria), and hemi-inattention (neglect).
Proportion of subjects with ≥4 point increase in NIHSS score during hospitalisation | D1~ Day 10
  The NIHSS is a 15-item impairment scale, which provides a quantitative measure of key components of a standard neurological examination.
  The scale assesses level of consciousness, extraocular movements, visual fields, facial muscle function, extremity strength, sensory function, coordination (ataxia), language (aphasia), speech (dysarthria), and hemi-inattention (neglect).
Proportion of subjects with Barthel Index Scale (BI) scores ≥95 on day 90 | Day 90
  The BI is a scale that measures ten basic aspects of activity related to self-care and mobility. The normal score is 100, and lower scores indicate greater dependency.
Day 90 European Five Dimensional Health Scale (EQ-5D) Score | Day 90
  The EQ-5D is a generic HRQoL measurement with evidence of good reliability and validity in various disease populations, including stroke. The EQ-5D contains the self- reported health state profile of five dimensions (mobility, self-care, usual activity, pain/discomfort, and depression/ anxiety) and a visual analog scale (EQ-VAS) .
Mortality due to stroke within 90 days | Day 90
  Mortality due to stroke within 90 days
Change in infarct volume from baseline after 24 hours of dosing | 24 hours after treatment
  Change in infarct volume from baseline after 24 hours of dosing

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Harrison International Peace Hospital, Hengshui, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Anyang People's Hospital, Anyang, Henan
  - Nanshi Hospital of Nanyang, Nanyang, Henan
  - Nanyang Second General Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Nanyang Medicinal College, Nanyang, Henan
  - MeiHekou Central Hospital, Meihekou, Jilin
  - Beipiao Central Hospital, Chaoyang, Liaoning
  - Ceneral Hospital of Mining Industry Group Fuxin, Fuxin, Liaoning
  - The Affiliated Hospital of Shenyang Medical College, Shenyang, Liaoning
  - The First People's Hospital of Shenyang, Shenyang, Liaoning
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - Iron Coal General Hospital of Liaoning Health Industry Group, Tieling, Liaoning
  - Keshketengqi Hospital of Traditional Chinese Medicine and Mongolian Medicine, Chifeng, Neimenggu
  - Xianyang Hospital of Yan'an University, Xianyang, Shaanxi
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Tengzhou Central People's Hospital, Tengzhou, Shandong
  - Sinopharm Tongmei General Hospital, Datong, Shanxi
  - Linfen Central Hospital, Linfen, Shanxi
  - Linfen People's Hospital, Linfen, Shanxi
  - Beijing Tiantan Hospital , Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Undecided